CLINICAL TRIAL: NCT00922883
Title: A Pilot Study of a Thrombopoietin-Receptor Agonist (TPO-R Agonist), Eltrombopag, in Aplastic Anemia Patients With Immunosuppressive-Therapy Refractory Thrombocytopenia
Brief Title: A Pilot Study of the Thrombopoietin-Receptor Agonist Eltrombopag in Refractory Aplastic Anemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090154; 09-H-0154 (Other: The National Institutes of Health)
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Anemia, Aplastic; Anemia, Hypoplastic; Thrombocytopenia
Keywords: Promacta; SAA; Aplastic Anemia; Thrombocytopenia
MeSH Terms: conditions — Anemia, Aplastic; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental): Eltrombopag (Promacta): Subjects commenced eltrombopag at a dose of 50 mg, which was increased by 25 mg every 2 weeks if the platelet count had not increased by 20 × 103/µL, to a maximum dose of 150 mg.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag
  Other Names: Promacta

SUMMARY:
Severe aplastic anemia (SAA) is a life-threatening blood disease which can be effectively treated with immunosuppressive drug regimens or allogeneic stem cell transplantation. However, 20-40% of patients without transplant options do not respond to immunosuppressive therapies, and have persistent severe cytopenias, requiring regular platelet transfusions, which are expensive and inconvenient, and are a risk for further serious bleeding complications.

Thrombopoietin (TPO) is the principal endogenous regulator of platelet production and also stimulates hematopoietic stem and progenitor cells. A small molecule oral TPO-agonist, eltrombopag has been shown to increase platelets in healthy subjects and in patients with immune thrombocytopenic purpura (ITP), and received FDA approval in 2008 for the treatment of thrombocytopenia in ITP. This Phase 2, non-randomized pilot study of eltrombopag in aplastic anemia patients with immunosuppressive therapy refractory thrombocytopenia will test the safety and potential efficacy of eltrombopag treatment patients with refractory thrombocytopenia following immunosuppression for aplastic anemia.

Subjects will initiate study medication at an oral dose of 50 mg/day, which will be increased up to 150 mg/day as clinically indicated to the lowest dose that maintains a stable platelet count 20,000/(micro)L above baseline while maximizing tolerability. Response will be assessed at 3-4 months. Platelet response is defined as platelet count increases to 20,000/L above baseline at three months. or stable platelet counts with transfusion independence for a minimum of 8 weeks. Erythroid response for subjects with a pretreatment hemoglobin of less than 9 g/dL will be defined as an increase in hemoglobin by greater than or equal to 1.5g/dL without packed red blood cell (PRBC) transfusion support, or a reduction in the units of transfusions by an absolute number of at least 4 PRBC transfusions for eight consecutive weeks compared with the pretreatment transfusion number in the previous 8 weeks. Neutrophil response will be defined in those with a pretreatment absolute neutrophil count (ANC) of less than 0.5 times 10(9)/L as at least a 100 percent increase or an absolute increase greater than 0.5 times 10(9)/L. Subjects with response at 3-4 months may continue study medication (extended access) until they meet an off study criteria. The primary objective is to assess the safety and efficacy of the oral thrombopoietin receptor agonist (TPO-R agonist) eltrombopag in aplastic anemia patients with immunosuppressive-therapy refractory thrombocytopenia. Secondary objectives include the analysis of the incidence and severity of bleeding episodes, and the impact on quality of life.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a life-threatening blood disease which can be effectively treated with immunosuppressive drug regimens or allogeneic stem cell transplantation. However, 20-40% of patients without transplant options do not respond to immunosuppressive therapies, and have persistent severe thrombocytopenia. Even patients that respond to immunosuppressive therapies with an improvement in their life-threatening neutropenia sometimes have persistent thrombocytopenia. Both groups of patients (i.e. nonresponders to immunosuppressive therapy and responders with persistent thrombocytopenia) require regular platelet transfusions, which are expensive and inconvenient, and are a risk for further serious bleeding complications.

Thrombopoietin (TPO) is the principal endogenous regulator of platelet production. On binding to the megakaryocyte progenitor TPO receptor, TPO initiates a number of signal transduction events to increase the production of mature megakaryocytes and platelets. Thrombopoietin also has stimulatory effects on more primitive multilineage progenitors and stem cells in vitro and in animal models. A 2nd generation small molecule TPO-agonist, eltrombopag (Promacta ) has been shown to increase platelets in healthy subjects and in thrombocytopenic patients with chronic immune thrombocytopenic purpura (ITP) and hepatitis C virus (HCV) infection. Eltrombopag is administered orally and has been well-tolerated in clinical trials. Unlike recombinant TPO, it has not been found to induce autoantibodies. Eltrombopag received FDA accelerated approval on Nov 20, 2008 for the treatment of thrombocytopenia in patients with chronic immune (idiopathic) thrombocytopenic purpura who have had an insufficient response to corticosteroids, immunoglobulins, or splenectomy.

Because a paucity of megakaryocytes and decreased platelet production is responsible for thrombocytopenia in aplastic anemia patients, we now propose this Phase 2, non-randomized pilot study of eltrombopag in aplastic anemia patients with immunosuppressive therapy refractory thrombocytopenia.

Subjects will initiate study medication at an oral dose of 50 mg/day (25 mg/day for East Asians), which will be increased or decreased as clinically indicated to the lowest dose that maintains a stable platelet count greater than or equal to 20,000/microL above baseline while maximizing tolerability. Platelet treatment response is defined as platelet count increases to 20,000/microL above baseline at three months, or stable platelet counts with transfusion independence for a minimum of 8 weeks. Erythroid response for subjects with a pretreatment hemoglobin of less than 9 g/dL will be defined as an increase in hemoglobin by greater than or equal to 1.5g/dL without packed red blood cell (PRBC) transfusion support, or a reduction in the units of transfusions by an absolute number of at least 4 PRBC transfusions for eight consecutive weeks compared with the pretreatment transfusion number in the previous 8 weeks. Neutrophil response will be defined in those with a pretreatment absolute neutrophil count (ANC) of less than 0.5 times 10(9)/L as at least a 100 percent increase or an absolute increase greater than 0.5 times 10(9)/L. Subjects with a platelet, erythroid, and/or neutrophil response at 12 weeks may continue study medication (extended access) until they meet an off study criteria. Subjects with platelet, erythroid, or neutrophil response at 12 weeks may continue study medication for an additional 4 weeks (to ensure eligibility) prior to being consented for entry into the extended access part of the trial. Patients may remain on the extended access trial until they met an off study criteria.

The primary objective is to assess the safety and efficacy of the oral thrombopoietin receptor agonist (TPO-R agonist) eltrombopag in aplastic anemia patients with immunosuppressive-therapy refractory thrombocytopenia.

Secondary objectives include the analysis of the incidence and severity of bleeding episodes, and the impact on quality of life.

The primary endpoint will be the portion of drug responders as defined by changes in the platelet count and/or platelet transfusion requirements, hemoglobin levels, number of red blood cell transfusions, or neutrophil counts as measured by International Working Group criteria and the toxicity profile as measured using the CTCAE criteria. Platelet treatment response is defined as platelet count increases to 20,000/microL above baseline at three months, or stable platelet counts with transfusion independence for a minimum of 8 weeks. Erythroid response for subjects with a pretreatment hemoglobin of less than 9g/dL will be defined as an increase in hemoglobin by greater than or equal to 1.5g/dL or a reduction in the units of PRBC transfusions by at least 50% during the eight consecutive weeks prior to response assessment compared with the pretreatment transfusion number in the previous 8 weeks. Neutrophil response will be defined in those with pretreatment absolute neutrophil count (ANC) of less than 0.5 times 10(9)/L as at least a 100 percent increase in ANC, or an ANC increase greater than 0.5 times 10(9)/L.

Secondary endpoints will include incidence of bleeding; changes in serum thrombopoietin level (as measured by enzyme-linked immunosorbent assay, R&D Systems), and health related quality of life (as measured by the Medical Outcomes Study 36-Item Short Form General Health Survey, version 2 [SF36v2J]; Quality-Metric) measured at 12 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosis of aplastic anemia, with refractory thrombocytopenia following at least one treatment course of horse or rabbit ATG/cyclosporine.
  2. Platelet count less than or equal to 30,000/microL
  3. Age greater than or equal to 12 years old

EXCLUSION CRITERIA:

1. Diagnosis of Fanconi anemia
2. Infection not adequately responding to appropriate therapy
3. Patients with a PNH clone size in neutrophils of greater than or equal to 50%
4. HIV positivity
5. Creatinine > 2.5
6. Bilirubin > 2.0
7. SGOT or SGPT > 5 times the upper limit of normal
8. Hypersensitivity to eltrombopag or its components
9. Female subjects who are nursing or pregnant or are unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential
10. History of malignancy other than localized tumors diagnosed more than one year previously and treated surgically with curative intent (for instance squamous cell or other skin cancers, stage 1 breast cancer, cervical carcinoma in situ, etc)
11. Unable to understand the investigational nature of the study or give informed consent
12. History of congestive heart failure arrhythmia requiring chronic treatment, arterial or venous thrombosis (not excluding line thrombosis) within the last 1 year, or myocardial infarction within 3 months before enrollment
13. ECOG Performance Status of 3 or greater
14. Treatment with horse or rabbit ATG or Campath within 6 months of study entry. Concurrent stable treatment with cyclosporine or G-CSF is permitted.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-05-29; Primary Completion 2013-05-07 (Actual); Study Completion 2018-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia E Dunbar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS, Calado RT, Scheinberg P. Current concepts in the pathophysiology and treatment of aplastic anemia. Blood. 2006 Oct 15;108(8):2509-19. doi: 10.1182/blood-2006-03-010777. Epub 2006 Jun 15. PMID 16778145
- [Background] Emmons RV, Reid DM, Cohen RL, Meng G, Young NS, Dunbar CE, Shulman NR. Human thrombopoietin levels are high when thrombocytopenia is due to megakaryocyte deficiency and low when due to increased platelet destruction. Blood. 1996 May 15;87(10):4068-71. PMID 8639762
- [Result] Desmond R, Townsley DM, Dumitriu B, Olnes MJ, Scheinberg P, Bevans M, Parikh AR, Broder K, Calvo KR, Wu CO, Young NS, Dunbar CE. Eltrombopag restores trilineage hematopoiesis in refractory severe aplastic anemia that can be sustained on discontinuation of drug. Blood. 2014 Mar 20;123(12):1818-25. doi: 10.1182/blood-2013-10-534743. Epub 2013 Dec 17. PMID 24345753
- [Result] Olnes MJ, Scheinberg P, Calvo KR, Desmond R, Tang Y, Dumitriu B, Parikh AR, Soto S, Biancotto A, Feng X, Lozier J, Wu CO, Young NS, Dunbar CE. Eltrombopag and improved hematopoiesis in refractory aplastic anemia. N Engl J Med. 2012 Jul 5;367(1):11-9. doi: 10.1056/NEJMoa1200931. PMID 22762314
- [Derived] Winkler T, Fan X, Cooper J, Desmond R, Young DJ, Townsley DM, Scheinberg P, Grasmeder S, Larochelle A, Desierto M, Valdez J, Lotter J, Wu C, Shalhoub RN, Calvo KR, Young NS, Dunbar CE. Treatment optimization and genomic outcomes in refractory severe aplastic anemia treated with eltrombopag. Blood. 2019 Jun 13;133(24):2575-2585. doi: 10.1182/blood.2019000478. Epub 2019 Apr 16. PMID 30992268
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-H-0154.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 patients were consented, but 1 patient was removed before treatment with the investigational agent was initiated because an additional review of baseline bone marrow revealed that the patient was not eligible, because the patient had changes in the bone marrow inconsistent with a diagnosis of aplastic anemia.
Period: Overall Study
Arm/Group | Eltrombopag
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Note that baseline information was available on the 44 patients consented and enrolled, but one patient was removed from protocol before initiation of the investigative agent, and thus adverse events and results information refers only to 43 patients
Arm/Group | Eltrombopag
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 27
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 21
  More than one race | 3
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: The Portion of Drug Responders as Defined by Hematologic Improvements
Description: Defined as unilineage or multilineage recovery by 1 or more of the following: 1) platelet response (increase to 20 × 103/μL above baseline or stable platelet counts with transfusion independence for a minimum of 8 weeks in those who were transfusion dependent on entry into the protocol); (2) erythroid response (when pretreatment hemoglobin was <9 g/dL, defined as an increase in hemoglobin by 1.5 g/dL or, in transfused patients, a reduction in the units of packed red blood cell transfusions by an absolute number of at least 4 transfusions for 8 consecutive weeks, compared with the pretreatment transfusion number in the previous 8 weeks); and (3) neutrophil response (when pretreatment absolute neutrophil count [ANC] of <0.5 × 103/μL as at least a 100% increase in ANC, or an ANC increase >0.5 × 103/μL, and the toxicity profile as measured using Common Terminology Criteria for Adverse Events).
Time Frame: 12-16 weeks
Population: All subjects who received Eltrombopag were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 43
Participants | 17

ADVERSE EVENTS:
Arm/Group | Eltrombopag
All-Cause Mortality (participants affected / at risk) | 4/43
Serious Adverse Events (participants affected / at risk) | 16/43
Other Adverse Events (participants affected / at risk) | 38/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=43)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Clostridium difficile colitis (Gastrointestinal disorders) | 1
Gingivitis ulcerative (Gastrointestinal disorders) | 1
Drug eruption (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic neoplasm (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=43)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 1
Jaundice (Blood and lymphatic system disorders) | 1
Petechiae (Blood and lymphatic system disorders) | 3
Purpura (Blood and lymphatic system disorders) | 1
Chest pain (Cardiac disorders) | 2
Dizziness (Cardiac disorders) | 4
Dyspnoea (Cardiac disorders) | 1
Dyspnoea exertional (Cardiac disorders) | 2
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 2
Dry eye (Eye disorders) | 2
Eye contusion (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Myopia (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal injury (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Anal fissure (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 2
Gingival disorder (Gastrointestinal disorders) | 1
Gingival swelling (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Oral candidiasis (Gastrointestinal disorders) | 1
Oropharyngeal pain (Gastrointestinal disorders) | 4
Pelvic organ injury (Gastrointestinal disorders) | 1
Pericoronitis (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Tooth abscess (Gastrointestinal disorders) | 1
Tooth injury (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Axillary pain (General disorders) | 1
Catheter site pain (General disorders) | 1
Fatigue (General disorders) | 11
Induration (General disorders) | 1
Injection site infection (General disorders) | 1
Night sweats (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 1
Hepatitis viral (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Rhinitis allergic (Immune system disorders) | 2
Urticaria (Immune system disorders) | 2
Cellulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 8
Viral infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 1
Osteoporosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Piriformis syndrome (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 7
Insomnia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Personality disorder (Psychiatric disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Platelet transfusion (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Haematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes